CLINICAL TRIAL: NCT02064452
Title: Evaluating an Online Parenting Support System Disseminated by Pediatric Practices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DA021307-06A1; 2R01DA021307-06A1 (NIH)
Record Dates: First submitted 2014-02-12; First posted 2014-02-17 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Child Disruptive Behavior Disorders; Oppositional Defiant Disorder; Conduct Disorder; Attention Deficit Hyperactivity Disorder
Keywords: behavior problems; children; prevention; parenting; online; pediatric
MeSH Terms: conditions — Oppositional Defiant Disorder; Conduct Disorder; Attention Deficit Disorder with Hyperactivity; Mental Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Triple P Online System (Experimental): The Triple P Online System (TPOS) is an interactive, video-driven online parenting support website, delivered with 3 different levels of intensity, depending on severity of children's behavior problems. In this arm, pediatric clinics are randomized to receive training in child disruptive behavior disorders, Triple P principles and target parenting strategies, the Triple P Online System, effectively referring eligible families to TPOS, and supporting their use of the program. Referred parents in this condition receive access to TPOS immediately.
  Interventions: Other: Triple P Online System
- Enhanced Usual Community Care-Waitlist (Placebo Comparator): In this arm, pediatric clinics are randomized to receive access for their parents and practitioners to a referral website designed to assist parents of children with disruptive behavior disorders in accessing appropriate community resources; on the website, community resources for treatment of child disruptive behavior disorders (mental health services, parenting services) are described and can be searched by location, cost, and acceptance of Medicare. Parents in this condition receive access to the Triple P Online System (TPOS) after completion of their 1-year follow-up assessment. Pediatricians receive free training in TPOS at the end of their waiting period.
  Interventions: Behavioral: Placebo Comparator

INTERVENTIONS:
Other: Triple P Online System — The Triple P Online System (TPOS) is an online parenting support program designed to assist parents in developing effective parenting practices for handling their children's problem behaviors. Content focuses on positive attention and praise, teaching strategies, effective discipline, antecedent strategies to avoid problems in high-risk situations, and applying these principles to specific situations. TPOS integrates 3 different levels of program intensity to meet different levels of family need, based on severity of children's behavior problems.
  Arms: Triple P Online System
Behavioral: Placebo Comparator — Enhanced Usual Community Care-Waitlist
  Arms: Enhanced Usual Community Care-Waitlist

SUMMARY:
This study will experimentally evaluate an internet-based version of the Triple P Positive Parenting Program, the Triple P Online System (TPOS), which presents the Triple P content in an interactive, video-enriched, and personalized format with 3-levels of flexible dosage, and will compare it against usual community services. Thirty pediatric clinics involving 100 practitioners in 9 counties across western Washington will be recruited and randomized to receive (a) access for their patients to the Triple P Online System and training in how to effectively promote TPOS and advise parents on their children's behavior problems or (b) Usual Care Community-Waitlist Control, in which parents will be assisted with an appropriate referral for services in the community.

DETAILED DESCRIPTION:
Disruptive behavior problems are among the most prevalent mental health conditions for young children, and they carry significant risks for later socioemotional, conduct, and academic problems, such as substance abuse, delinquency, and school failure. How parents handle these challenging behaviors strongly influences their children's long-term trajectory. Evidence-based parenting programs have shown much value in reducing early-onset disruptive behavior problems, thereby reducing risks for later substance abuse and other behavioral health problems. The reach of parenting programs is limited, however, by significant challenges in recruiting, engaging, and retaining parents, such that most parents who could benefit from parenting assistance never receive it. A public health approach for improving parenting practices that makes evidence-based parenting programs widely available and accessible in a range of formats could reduce the prevalence of disruptive behavior problems, and thus the population-level risk for substance abuse and other adverse outcomes. Internet-based intervention offers significant potential as part of a population-wide strategy for bringing evidence-based parenting practices to a broad range of parents experiencing challenges in raising their children. Furthermore, pediatricians could be a natural touchpoint for reaching families with evidence-based parenting supports. The field knows little, however, about the potential of the internet to strengthen parenting practices, or about how pediatric practitioners might be engaged in improving the reach of an online parenting program. This study will experimentally evaluate an internet-based version of the Triple P Positive Parenting Program, the Triple P Online System (TPOS), which presents the Triple P content in an interactive, video-enriched, and personalized format with 3-levels of flexible dosage, and will compare it against usual community services. Thirty pediatric clinics involving 100 practitioners in 9 counties across western Washington will be recruited and randomized to receive (a) access for their patients to the Triple P Online System and training in how to effectively promote TPOS and advise parents on their children's behavior problems or (b) Usual Care Community-Waitlist Control, in which parents will be assisted with an appropriate referral for services in the community. Practitioners will recruit into their respective conditions 400 families of 3-8 year-old children with elevated behavior problems. Measures of parents' parenting practices, family functioning, children's disruptive behavior problems, and practitioners' protocols for advising on behavior problems will be obtained at baseline, post-intervention, and 1-year follow-up. The efficacy of the Triple P Online System in improving these outcomes will be examined, as well as dosage-response relationships. This study will further our understanding of the potential value of promoting internet-based parenting programs through pediatric practitioners. Maximizing the reach of evidence-based parenting programs has the potential to reduce the prevalence of children's behavior problems, and thus reduce risks for later problems such as substance abuse.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric practitioners at participating clinics in western Washington.
* Families of children 3-8 years old referred by participating pediatric practitioners. Eligible families will: (a) have a child 3-8 years old, (b) have at least half-time custody of the child, (c) care for the child at least 16 waking hours per week, (d) express concern to their practitioner about difficulties with the child's behavior, (e) score .80 standard deviation or more above the normed mean on the Eyberg Child Behavior Inventory, (f) speak English, and (g) have regular access to high-speed internet.

Exclusion Criteria:

* None.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2014-05 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Change from Baseline at T2 and T3 on Parenting and Family Adjustment Scale (Sanders & Morawska, 2010) | T1 (Baseline), T2 (16 weeks after T1), T3 (1 year after T2).
  40-item parent-report questionnaire; assesses discipline practices, positive parenting, parent mood, family relationships, and co-parenting support at T1 (Baseline), T2 (16 weeks after T1), T3 (1 year after T2).

SECONDARY OUTCOMES:
Child Adjustment and Parent Efficacy Scale (Morawska & Sanders, 2010) | T1 (Baseline), T2 (16 weeks after T1), T3 (1 year after T2).
  Parent-report questionnaire; 30 items measure children's emotional and behavioral problems and positive behaviors; 20 items measures parents' self-efficacy for handling the problem behaviors
Knowledge of Effective Parenting Scale (Winter, Morawska, & Sanders, 2011) | T1 (Baseline), T2 (16 weeks after T1), T3 (1 year after T2).
  Multiple-choice parenting knowledge quiz
Child and Adolescent Disruptive Behavior Inventory (Burns, Taylor, & Rusby, 2001) | T1 (Baseline), T2 (16 weeks after T1), T3 (1 year after T2).
  Parent-report questionnaire measuring children's oppositional behavior to adults, oppositional behavior to other children, hyperactivity, and conduct problems
Parent Daily Report (adapted from Chamberlain & Reid, 1987), coded with the Parent Discipline Interview Coding System (Rusby, Metzler, Sanders & Ware, 2010) | T1 (Baseline), T2 (16 weeks after T1), T3 (1 year after T2).
  Series of 3 phone interviews with mother at each timepoint; mother reports on frequency of specific problematic and positive child behaviors over the past 24 hours. Mother reports how she handled the two most problematic behaviors; answers are coded by independent coders.
Preschool Age Psychiatric Assessment (Egger & Angold, 2004) | T1 (Baseline), T3 (1 year after T2).
  Diagnostic interview, administered over the phone to mothers, used for study children ages 3-5; modules assessing Oppositional Defiant Disorder, Conduct Disorder, and Attention Deficit Hyperactivity Disorder are utilized.
National Institute of Mental Health Diagnostic Interview Schedule for Children Version IV (Shaffer, Fisher, Lucas, Dulcan & Schwab-Stone, 2000) | T1 (Baseline), T3 (1 year after T2).
  Diagnostic interview, administered over the phone to mothers, used for study children ages 6-8; modules assessing Oppositional Defiant Disorder, Conduct Disorder, and Attention Deficit Hyperactivity Disorder are utilized.
Pediatricians' self-efficacy for advising parents of children with conduct problems, typical referral patterns for these problems, attitudes toward evidence-based self-administered parenting interventions | T1 (Baseline), T2 (10 months after T1), T3 (1 year after T2).
  pediatrician-reported questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Carol W Metzler, PhD, Principal Investigator — Oregon Research Institute
Locations (2):
- United States (2):
  - Oregon Research Institute, Eugene, Oregon
  - Seattle Children's Research Institute, Seattle, Washington